CLINICAL TRIAL: NCT04291482
Title: A Theory-based Digital Intervention to Promote Weight Loss and Weight Loss Maintenance (Choosing Health): A Randomised Controlled Trial With Within Person Assessment
Brief Title: A Theory-based Digital Intervention to Promote Weight Loss and Weight Loss Maintenance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: POIR.04.04.00-00-5CF3/18-00
Record Dates: First submitted 2020-02-04; First posted 2020-03-02 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Overweight and Obesity
Keywords: Diet; Physical activity; Behaviour change; Behaviour maintenance; Weight loss; Within-person design; Digital health
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Weight Loss

STUDY DESIGN:
Intervention Model Description: This is a two-group intervention trial adopting a randomised controlled design. It is a hybrid trial assessing intervention effectiveness, cost-effectiveness and implementation with embedded within person assessment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and Outcomes Assessor will be blinded to participants study arm allocation. It is impossible to blind study participants and intervention providers, it is behavioural trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The intervention group participants will be assessed with EMA and they will provide daily data regarding their predictors of weight loss outcomes and their adherence to the personal weight loss plan (phase I, month 0-3). Then participants will receive tailored information regarding the most predictive factors relevant to their weight loss trajectories (phase II, month 3-6). The information will be tailored and delivered through emails and text messages.
  Interventions: Behavioral: Choosing Health Intervention
- Control arm (Other): Control group participants will receive basic educational weight loss information in a form of educational factual emails and text messages.
  Interventions: Behavioral: Choosing Health Control

INTERVENTIONS:
Behavioral: Choosing Health Intervention — The intervention consists of information materials provided at baseline in a form of eBook or a physical book depending on participants preferences. The book includes the rationale for the intervention, basic information on healthy eating and behaviour change and tables allowing self-monitoring of weight, physical activity and eating (i.e., brief food diary). The book is non-tailored and it has weekly tasks for the participants to complete during 26 weeks (initial 6 months) to support their weight loss. The intervention group will also receive a series of daily text messages and weekly email messages supporting their weight loss and promoting weight loss maintenance. In phase I (month 0-3), the messages and emails will be generic and factual; in the phase II of the intervention, participants will receive text messages and emails tailored to the strongest predictors of outcomes identified in phase I.
  Arms: Intervention arm
Behavioral: Choosing Health Control — The control consists of information materials provided at baseline in a form of eBook or a physical book depending on participants preferences. The book includes the rationale for the intervention and basic information on healthy eating and physical activity. The control group will also receive monthly email messages with generic and factual information.
  Arms: Control arm

SUMMARY:
Obesity can severely reduce quality and longevity of life and there is an urgent need to help people lose weight and maintain weight loss long term. Digital behaviour change interventions targeting diet and physical activity have the potential for public health gain; however, these interventions are often not adequately tailored to the participants. The aim of this study is to develop and test a digital intervention to help people make sustainable changes to diet and physical activity, and consequently their weight. This study is a hybrid trial that will evaluate the effectiveness, cost-effectiveness and implementation of the Choosing Health program among overweight/obese adults.

This study is a two-group randomised controlled trial (RCT) with within person assessment. Participants (N=285) will be randomly assigned to either the Choosing Health digital intervention or a control group. For intervention participants, Ecological Momentary Assessment (EMA) will be used to identify behavioural determinants for each individual in order to tailor evidence-based behaviour change techniques and intervention content. Control group will receive non-tailored factual weight loss advice. Primary outcome is mean difference in weight loss between groups at 6 months, in kilograms. Key outcomes will be measured at baseline, 3-, 6- and 12 months. Data will be analysed using multilevel modelling and time series analysis.

This is the first weight loss intervention applying individualised digital tailoring based on continuous assessment of individual's psychological determinants of behaviour measured over time. The Choosing Health will offer insight into factors associated with success in making sustained changes to weight, and secondary outcomes, such as diet and physical activity.

DETAILED DESCRIPTION:
Behavioural science offers theory-driven and evidence-based behaviour change techniques that can support people in losing weight and maintaining it long term. These techniques have not yet been assessed in within-person studies that not only examine aggregated between-group effects (e.g., intervention versus control comparisons) but also determine personal trajectories of weight loss and maintenance and tailor accordingly to the strongest predictors of outcomes. The aim of the proposed study is to develop and test a digital intervention that uses Ecological Momentary Assessment (EMA) and tailors the evidence-based behaviour change techniques that are based on theory to the strongest predictors of outcomes (based on EMA responses collected over time).

This study will determine the effectiveness and cost-effectiveness of the proposed intervention through the Randomised Controlled Trial (EMA tailored intervention versus control), with within person component embedded in the trial. Study hypothesis is that participants in the EMA tailored intervention group will lose significantly more weight than participants in the control group from baseline to 6 months (post program comparison - primary outcome) and at 12 months (maintenance effects assessment - secondary outcome).

This is a two-group intervention trial adopting a randomised controlled design. It is a hybrid trial assessing intervention effectiveness, cost-effectiveness and implementation. This study has within person component embedded in the design and intervention group will answer EMA questions during the initial 3 months of the study and will receive tailored intervention at month 3 combined with additional EMA. There are two phases of the 6-month intervention (I) observational EMA phase and (II) active intervention phase.

The proposed intervention is delivered online through emails and text messages and based on the EMA responses in phase I, it is tailored in phase II. The intervention will have a non-automatic component, meaning trained facilitators will answer participants' queries and provide additional resources if and when needed to improve the engagement with the intervention. The study meets CONSORT criteria for RCTs and study ethical approval was obtained from SWPS University of Social Sciences and Humanities, Wroclaw, Poland (approval number 03/P/12/2019).

ELIGIBILITY:
Inclusion Criteria:

* Adults with overweight and obesity (18+);
* Individuals with a BMI 25 and higher at the baseline assessment.

Exclusion Criteria:

* Individuals who self-report a physical condition or impairment preventing them from being physically active or losing excess body weight;
* Individuals who have had a bariatric surgery or are planning to have one within the next 12 months;
* Individuals who are currently participating in another weight loss program (e.g., regular meetings with personal trainer);
* Individuals who report any contradictions to exercise as indicated by the PAR-Q or pregnant women who consulted their doctor to obtain approval to take part in the study and did not get the approval;
* Individuals who do not have a mobile phone with access to the internet;
* Individuals who are currently participating in another weight loss program (e.g., regular meetings with personal trainer);
* Pregnant women;
* Individuals who are planning to move outside of the study region and are not willing to travel for study measurement sessions;
* Individuals who are on medication that causes weight gain;
* Individuals with a pacemaker (the scale used in the study is not appropriate for use in these individuals).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight | Change from baseline to 6 months
  Mean difference in weight loss between groups at 6 months, in kilograms

SECONDARY OUTCOMES:
Weight | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Objective measures of weight in kilograms
Height | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Objective measures of height in centimetres
BMI | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Weight and height will be combined to report BMI in kg/m^2
Body fat % | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Objective measures of body fat %
Systolic and diastolic blood pressure | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Objective measures of systolic and diastolic blood pressure measured in units of millimeters of mercury (mmHg)
Diet | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Measured with the Dietary Instrument for Nutrition Education (fatty foods, fruit and vegetable, and sugary food consumption). High scores are indicative of high consumption. Higher scores for fruit and vegetable mean a better outcome (0-3 scale; 1 item) and higher scores for fatty foods (0-24; 8 items on 0-3 scale) and sugary food (0-9; 3 items on 0-3 scale) mean a worse outcome. The minimum values are 0 and the maximum values are specified above in brackets.
Alcohol | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Measured with the Audit C; scale 0-12, high scores are indicative of high consumption.
Physical activity (self-reported) and sitting time | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Measured with the International Physical Activity Questionnaire short version, the minimum value is 0 (no activity), higher scores mean a better outcome. All activity will be converted to minutes before calculating MET minutes (total score). In each category a maximum of 21 hours of activity are permitted a week (3 hours X 7 days). To calculate MET minutes a week the MET value given (walking = 3.3, moderate activity = 4, vigorous activity = 8) will be multiplied by the minutes the activity was carried out and again by the number of days that that activity was undertaken. To get total MET minutes of physical activity a week the MET minutes achieved in each category (walking, moderate activity and vigorous activity) will be added.
Sleep duration and quality | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Measured with the Pittsburgh Sleep Quality Index. In scoring the Pittsburgh Sleep Quality Index, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Health related quality of life | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Measured with the EQ-5D-5 L (this is the unabbreviated scale title), the scale has five domains each scored on 1-5 scale; min 5 maximum 25 for all domains combined) higher scores mean a worse outcome and visual analogue scale is the second part of the questionnaire, asking to mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100. There are notes at the both ends of the scale that the bottom rate (0) corresponds to " the worst health you can imagine", and the highest rate (100) corresponds to "the best health you can imagine".
Number of adverse effects | Through study completion, an average of 1 year
  report of any adverse effects that may occur during the intervention
Self-reported measures of intentions | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Theory-derived psychological construct measured with 2 items addressing intentions (1-5 scale), the minimum and maximum values for the scale are 2-10, and higher scores mean a better outcome (higher intentions).
Self-reported measures of motivation | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Theory-derived psychological construct measured with 2 items addressing motivation (1-5 scale), the minimum and maximum values for the scale are 2-10, and higher scores mean a better outcome (higher motivation).
Self-reported measures of self-efficacy | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Theory-derived psychological construct measured with 2 items addressing self-efficacy (1-5 scale), the minimum and maximum values for the scale are 2-10, and higher scores mean a better outcome (higher self-efficacy).
Self-reported measures of attitudes | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Theory-derived psychological construct measured with 2 items addressing attitudes (1-5 scale), the minimum and maximum values for the scale are 2-10, and higher scores mean a better outcome (higher attitudes).
Self-reported measures of action planning | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Theory-derived psychological construct measured with 8 items addressing action planning (1-5 scale), the minimum and maximum values for the scale are 8-40, and higher scores mean a better outcome (better action planning).
Self-reported measures of coping planning | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Theory-derived psychological construct measured with 6 items addressing action planning (1-5 scale), the minimum and maximum values for the scale are 6-30, and higher scores mean a better outcome (better coping planning).
Self-reported measures of goal facilitation | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Theory-derived psychological construct measured with 2 items addressing goal facilitation (1-5 scale), the minimum and maximum values for the scale are 2-10, and higher scores mean a better outcome (better goal facilitation)
Self-reported measures of goal conflict | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Theory-derived psychological construct measured with 2 items addressing goal conflict (1-5 scale), the minimum and maximum values for the scale are 2-10, and higher scores mean a worse outcome (higher goal conflict)
Self-reported measures of habit strength for physical activity | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Theory-derived psychological construct measured with h self-report behavioural automaticity index for physical activity, 4 items (1-5 scale); the minimum and maximum values for the scale are 4-20, and higher scores mean a better outcome (habit strength)
Self-reported measures of habit strength for healthy eating | baseline (Time 0), 3 months (Time 1), 6 months (Time 2) and 12 months (Time 3)
  Theory-derived psychological construct measured with self-report behavioural automaticity index for healthy eating, 4 items (1-5 scale); the minimum and maximum values for the scale are 4-20, and higher scores mean a better outcome (habit strength)

OTHER OUTCOMES:
Demographic variables | baseline (Time 0)
  Age, sex, marital status, ethnicity, education, height (to calculate BMI), and household income

CONTACTS AND LOCATIONS:
Overall Officials: Felix Naughton, PhD, Principal Investigator — University of East Anglia; Aleksandra Luszczynska, Prof, Principal Investigator — SWPS University of Social Sciences and Humanities; Dominika Kwasnicka, PhD, Principal Investigator — SWPS University of Social Sciences and Humanities; Martin Hagger, Prof, Principal Investigator — University of California; Eleanor Quested, PhD, Principal Investigator — Curtin University
Locations (1):
- SWPS University, Wroclaw, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
We will share anonymised data using Open Science Framework.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available on the OSF after the study is completed.
Access Criteria: Anonymised data will be publicly available to access through the OSF.

REFERENCES:
- [Derived] Kwasnicka D, Luszczynska A, Hagger MS, Quested E, Pagoto SL, Verboon P, Robinson S, Januszewicz A, Idziak P, Palacz I, Naughton F. Theory-based digital intervention to promote weight loss and weight loss maintenance (Choosing Health): protocol for a randomised controlled trial. BMJ Open. 2020 Nov 23;10(11):e040183. doi: 10.1136/bmjopen-2020-040183. PMID 33234638
- See also: Study website — http://www.wybieramyzdrowie.pl/